CLINICAL TRIAL: NCT03962205
Title: Promoting Weight Loss and Psychological Well-being in Obese Patients: Combination of Behavioral Life Style and Well-Being Intervention
Brief Title: Promoting Weight Loss and Psychological Well-being in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Chiara Rafanelli, Ordinary Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PWlPwb-OB
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: obese patients; psychological well being; weight loss; depression; psychological distress; life-style intervention; demoralization
MeSH Terms: conditions — Obesity; Psychological Well-Being; Weight Loss; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral life-style and well-being intervention (Experimental): Participants will receive 12 group-based 2-hour weekly sessions for life-style modification and then 4 group-based 2-hour weekly sessions of the well-being intervention in addition to the treatment as usual.
  Interventions: Behavioral: cognitive-behavioral life style intervention; Behavioral: wellbeing intervention; Other: treatment as usual
- Cognitive Behavioral life-style intervention (Placebo Comparator): Participants will receive 12 group-based 2-hour weekly sessions for life-style modification in addition to the treatment as usual.
  Interventions: Behavioral: cognitive-behavioral life style intervention; Other: treatment as usual

INTERVENTIONS:
Behavioral: cognitive-behavioral life style intervention — Cognitive Behavioral life-style modification: The intervention will be composed of 12 weekly sessions. Each session will last about two hours and will be administered in a group setting (maximum 20 participants). During the first two sessions, a clinician will introduce the program to the participants and motivate them to make life-style changes.In the next eight sessions a dietician will provide participants with basics of nutrition and will coach them to use a structured diary to monitor their eating behavior and physical activity. Next, a physician will introduce to the patients various weight loss surgeries in terms of the adverse events, indications and effects of each option.The last session will be held by a psychologist and will focus on providing participants with useful strategies to promote healthy eating habits and physical activity, including problem solving and goal setting.
Behavioral: wellbeing intervention — This program will consist of 4 weekly group-based sessions and each meeting will last about two hours. During the sessions, participants will be coached how to self-monitor their well-being episodes in everyday life, especially those associated with life-style change, by means of a structured diary. Patients will be then ecounraged to discuss their well-being experiences during group sessions, focusing on dysfunctional thoughts/beliefs interrupting them, fostering the identification of more functional thoughts. The psychologist will also teach them how to promote well-being situations through behavioral exercises and will introduce to the participants relevant psychological well-being dimensions (based on Carol Ryff's multidimensional model) associated with patients' experiences emerged during the treatment.
  Arms: Cognitive Behavioral life-style and well-being intervention
Other: treatment as usual — The treatment as usual will involve any recommendation given to the participants by their physicians, including diet, physical activity and medication.

SUMMARY:
The goal of the proposed research is to assess the effects of a sequential combination of lifestyle and well-being intervention on weight loss and psychological well-being. It is hypothesized that psychological well-being promotion as an adjunct to life-style intervention will outperform life style intervention alone in promoting weight loss and psychological well-being in obese individuals.

DETAILED DESCRIPTION:
The present study is a longitudinal, single blind, randomized controlled pilot trial. The participants will be recruited at the Center of Metabolism Diseases and Clinical Dietetics of Sant'Orsola Hospital in Bologna, directed by Prof. Giulio Marchesini Reggiani, after approval of the Ethics Committee of Azienda Ospedaliero-Universitaria of Bologna.

Patients attending the Center of Metabolism Diseases and Clinical Dietetics during the enrollment period will be screened for inclusion and exclusion criteria by care coordinators or clinicians. Eligible patients will be required to sign the informed consent form and the consent form for personal data processing. The researchers will be in charge of explaining the project to make sure that it is fully understood by the patients.

During the first 3 months, all the participants will undergo a behavioral program focusing on lifestyle modification. The participants who accomplish the program for life-style modification will be randomly assigned to either the control group or the experimental group. Generalized block randomization will be carried out by a computer program (the Random Allocation Software 2.0), with an allocation ratio of 1:1.

Participants in the experimental group will receive a four-session intervention on psychological well-being. Each session will last one hour and will be offered weekly, based on the principles of Well-Being Therapy. Patients in the control group will only receive a treatment as usual (TAU), according to the instructions given by their clinicians. Data will be collected for each participant through questionnaires and interviews at baseline, at the end of the life-style intervention, at the end of the well-being intervention, and at 6 months of follow-up after the intervention. Given the nature of this study, it will not be possible for participants and treatment delivers to be blinded. Trained researchers, masked to the experimental allocation of patients, will perform measurements and analyses of the data to minimize potential bias.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI ≥ 30)
* aged ≥18 years
* willing to participate in the study.

Exclusion Criteria:

* inability to provide informed consent to participate in the study (i.e. psychotic or mentally impaired patients);
* insufficient knowledge of Italian;
* presence of a medical condition associated with unintentional weight loss or gain;
* presence of major psychiatric illness and cognitive deficit;
* participation in another weight-loss program;
* use of medication for weight loss;
* history of weight loss surgery or weight loss surgery scheduled during the last year or within 16 months from the beginning of the study;
* being pregnant or intended pregnancy during the last year or within 16 months from the beginning of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
4-month Change in body weight in kg | Baseline, 4 months
  4-month average change in body weight (kg) from baseline to 4 months. Weight will be measured with a standard balance beam scale with the participant in a lightweight clothing.
4-month Change in body weight in % | Baseline, 4 months
  4-month average change in body weight as a percentage of start weight
10-month change in body weight in kg | Baseline, 10 months
  10-month average change in body weight (kg) from baseline to 10 months.
10-month change in body weight in % | Baseline, 10 months
  10-month average change in body weight as a percentage of start weight
16-month change in body weight in kg | Baseline, 16 months
  16-month average change in body weight (kg)
16-month change in body weight in % | Baseline, 16 months
  16-month average change in body weight as a percentage of start weight
Change in Body mass Index (BMI) | Baseline, 4 months,10 months,16 months
  It will be computed as body weight (kg) divided by the square of height (m²).

SECONDARY OUTCOMES:
Change in psychological well-being | Baseline, 4 months,10 months,16 months
  It will be measured with the Psychological WellBeing scale, a 42-item self-rating scale, which includes six dimensions: self-acceptance, positive relations with others, autonomy, environmental mastery, purpose in life and personal growth. The respondents are asked to indicate on a 6-likert scale the extent to which they agree with each statement. Each dimension may range from 7-42, with higher scores indicating greater psychological well-being.
Change in the prevalence of depression | Baseline, 4 months,10 months,16 months
  It will be measured by well-trained researcher with The Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders - 5th edition (SCID-5-CV).
Change in the prevalence of demoralization | Baseline, 4 months,10 months,16 months
  It will be measured by well-trained researchers with The Diagnostic Criteria for Psychosomatic Research-Revised Semi-Structured Interview- Revised (DCPR-R)
Change in psychological distress | Baseline, 4 months,10 months,16 months
  It will be measured by the Symptom Questionnaire (SQ), a 92-item self-rating instrument with dichotomous responses divided into 4 dimensions: depression, anxiety, somatization and hostility/irritability. Each dimension consists in a symptom sub-scale including 17 questions and a well being one with 6 questions. Scores may range from 0 to 17 for each symptom sub-scale and from 0 to 6 for each well-being sub-scale. For each dimension, higher scores indicate more severe psychological distress.
Change in lifestyle | Baseline, 4 months,10 months,16 months
  It will be measured with GOSPEL (GlObal Secondary Prevention strategiEs to Limit event recurrence after myocardial infarction - GOSPEL study) questionnaire, a 32-item self-rating instrument for the assessment of physical activity levels, eating habits, and stress levels used among patients who need to change their lifestyle.
  The subscale on physical activity includes eight 4-point items with a total score ranging from 0 (poor/absent physical activity) to 20 (very high physical activity).
  The subscale on eating habits consists of ten 4-point items regarding Mediterranean diet based on the frequency of healthy food consumption, with a total score ranging from 0 (worst) to 30 (best). Three additional 4-point items on eating behavior are also included: their total score may range from 0 (bad dietary behavior) to 9 (healthy dietary behavior).
  The subscale on stress management includes seven 4-point items which total score may range from 0 (inadequate) to 21 (optimal).

OTHER OUTCOMES:
Change in psychosocial profile | Baseline, 4 months,10 months,16 months
  It will be measured with the PsychoSocial Index (PSI). PSI is a 55-item self-rating scale, divided into 5 domains: 1) Sociodemographic and clinical data (12 questions on medical and demographic information); 2) Stress subscale (17 yes/no questions) with a score ranging from 0 to 17 (a higher score indicates greater stress); 3) Well-being subscale (6 yes/no questions) with a score ranging from 0 to 6 (a higher score indicates greater psychological well-being); 4) Psychological distress (15 four-point questions ranging from 0 to 3) with a total score from 0 to 45 (a higher score indicates greater psychological distress); 5) Abnormal Illness Behavior (3 four-point questions from 0 to 3) with a total score ranging from 0 to 9 (a higher score indicates more severe abnormal illness behavior). Finally, PSI includes one 4-point question on self-perceived quality of life, with a score from 0 to 4 (a higher score indicates better quality of life).
Change in motivation for weight change | Baseline, 4 months,10 months,16 months
  It will be measured by the Goal Related Weight Questionnaire (GRWQ), which asks the respondents to self-report their dream, happy, acceptable, and disappointed weight in kilograms in the first part (4 items) and to indicate to which extent they expect weight loss to impact various aspects of their psycho-social and health-related functioning, with each item scored from 1 (extremely negative) to 10 (extremely positive), in the second part (21 items).

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Rafanelli, MD,PhD, Study Director — University of Bologna
Locations (1):
- SSD Malattie del Metabolismo e Dietetica Clinica Policlinico Sant'Orsola- Malpighi, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fava GA. Well-Being Therapy: Current Indications and Emerging Perspectives. Psychother Psychosom. 2016;85(3):136-45. doi: 10.1159/000444114. Epub 2016 Apr 5. No abstract available. PMID 27043240